CLINICAL TRIAL: NCT07240688
Title: A Prospective Observational Study on the Association of Lingual Retraction With Hemodynamic Parameter Changes in Patients Receiving Dental Procedures Under General Anesthesia
Brief Title: Association Between Lingual Retraction and Hemodynamic Changes in Patients Receiving Dental Treatment Under General Anesthesia
Status: Recruiting | Type: Observational
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Gözde Nur Erkan, Assistant Professor, MD, Kırıkkale University
Other Study IDs: KU-ERKAN-003
Record Dates: First submitted 2025-11-14; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-10

CONDITIONS: Trigeminocardiac Reflex; Hemodynamic Changes; Dental Procedures
Keywords: Trigeminocardiac Reflex; Hemodynamic Changes; Lingual Retraction; Dental Procedures; General Anesthesia
MeSH Terms: conditions — Glossoptosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1. Pediatric Patients: Patients aged 0 to 17 years undergoing dental procedures under general anesthesia. No intervention beyond routine clinical care; observational monitoring of trigeminocardiac reflex and hemodynamic parameters.
- Group 2. Adult Patients: Patients aged 18 years and older undergoing dental procedures under general anesthesia. No intervention beyond routine clinical care; observational monitoring of trigeminocardiac reflex and hemodynamic parameters.

SUMMARY:
This study aims to investigate the association between sudden decreases in heart rate and blood pressure during dental procedures requiring lingual retraction-such as fillings, root canal treatments, tooth extractions, and cyst surgeries-under general anesthesia. Patients will be routinely monitored for vital parameters during anesthesia. Sudden drops in heart rate and blood pressure (10-20% decrease) will be recorded as lingual retraction-related trigeminocardiac reflex (TCR) events, along with the type of lingual retraction, dental procedure, and tooth location at the time of occurrence. Additionally, the results will be analyzed in relation to patient age, sex, and tongue size.

DETAILED DESCRIPTION:
Stimulation of both the central and peripheral branches of the trigeminal nerve can lead to clinically significant hemodynamic changes. The trigeminocardiac reflex (TCR), a brainstem-mediated reflex mechanism triggered by such stimulations, causes sudden and marked decreases in heart rate and arterial blood pressure. This reflex may result in hemodynamic instability during surgical interventions and, in rare cases, can precipitate severe cardiac complications including cardiac arrest.

While TCR is more commonly observed during ophthalmic, craniofacial, and skull base surgeries, it may also occur during dental procedures. Stimulation of the peripheral branches of the lingual nerve, such as during lingual retraction, has been associated with cardiovascular side effects like bradycardia. This phenomenon reflects systemic hemodynamic responses resulting from trigeminal nerve stimulation.

The literature reports significant drops in heart rate and arterial pressure due to TCR during common dental procedures such as tooth extraction and implant surgery. Notably, sudden decreases of 10-20% in blood pressure are considered clinically relevant indicators of TCR. Additionally, hemodynamic changes potentially related to this reflex have been documented during endodontic treatments, particularly in cases of irreversible pulpitis. Thus, stimulation of the dental branches of the trigeminal nerve may trigger TCR during dental procedures, leading to systemic hypotension.

In conclusion, TCR triggered by trigeminal nerve stimulation is an important hemodynamic reflex encountered during surgical and dental interventions. Early recognition and appropriate preventive measures are critical to mitigating potential cardiac risks. Clinical procedures should consider patients' susceptibility to such reflexes in planning and management.

This study aims to investigate the incidence of trigeminocardiac reflex triggered primarily by lingual retraction, and secondarily by dental procedure type, tooth location, patient age, and duration of general anesthesia in adult and pediatric patients undergoing dental surgeries under general anesthesia. Conducted at the operating rooms of Kırıkkale University Faculty of Dentistry, this prospective observational study will record TCR events using a specially designed patient monitoring form, correlating these events with various clinical factors.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to our faculty for dental procedures requiring general anesthesia.
* Patients classified as ASA physical status I or II.

Exclusion Criteria:

* Patients unwilling to participate in the study.
* Patients classified as ASA physical status III or IV.
* Patients with diseases affecting cardiac inotropy, chronotropy, or dromotropy.
* Patients using medications influencing cardiac inotropy, chronotropy, or dromotropy.
* Patients with cardiac pacemakers.
* Patients with cardiac arrhythmias.
* Patients with neurological disorders affecting the trigeminocardiac reflex pathway (inhibition or activation).

Ages: 2 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing dental procedures under general anesthesia at Kırıkkale University, Faculty of Dentistry, aged 2-65, classified as ASA physical status I or II. Both pediatric and adult patients will be included. Patients with cardiac or neurological conditions affecting the trigeminocardiac reflex will be excluded.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-10-13 (Actual); Primary Completion 2026-08-13 (Estimated); Study Completion 2026-10-13 (Estimated)

PRIMARY OUTCOMES:
Hemodynamic Changes Associated with Lingual Retraction | During the dental procedure (up to 4 hours)
  To quantify acute intraoperative alterations in heart rate and blood pressure related to lingual retraction during dental procedures performed under general anesthesia. Sudden decreases of ≥10-20% in these parameters will be defined and recorded as trigeminocardiac reflex (TCR) events.

SECONDARY OUTCOMES:
Incidence and Characteristics of TCR Events | During the dental procedure (up to 4 hours)
  To determine the overall incidence of lingual retraction-related TCR events and to characterize their severity and duration, including the magnitude of hemodynamic change and the need for pharmacologic or mechanical interventions.
Association of TCR Events With Procedural and Anatomic Factors | During the dental procedure (up to 4 hours)
  To evaluate the relationship between TCR occurrence and (a) the type of dental procedure (e.g., filling, root canal treatment, extraction, cyst surgery), (b) the method of lingual retraction, and (c) the treated tooth location (anterior/posterior; maxillary/mandibular).
Influence of Patient Characteristics on TCR Occurrence | During the dental procedure (up to 4 hours)
  To investigate the association between patient-specific factors-such as age, sex, and tongue size-and the likelihood of developing TCR during lingual retraction under general anesthesia.

CONTACTS AND LOCATIONS:
Locations (1):
- Kırıkkale University, Faculty of Dentistry, Kırıkkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be publicly available but may be shared upon reasonable request with qualified researchers, subject to approval by the study team and compliance with ethical and confidentiality guidelines.